CLINICAL TRIAL: NCT02671318
Title: Conversion to Sirolimus: Effects in Cytomegalovirus Infection Recurrence in Kidney Transplant Recipients (StopCMV: S=Sirolimus CMV= Cytomegalovirus)
Brief Title: Conversion to Sirolimus: Effects in Cytomegalovirus Infection Recurrence
Acronym: StopCMV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital do Rim e Hipertensão (Other)
Responsible Party: Principal Investigator, Geovana Basso, MD, Hospital do Rim e Hipertensão
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 43102815.0.0000.5505
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Cytomegalovirus Infections
Keywords: cytomegalovirus; sirolimus; cytomegalovirus recurrence; kidney transplant; conversion
MeSH Terms: conditions — Cytomegalovirus Infections | interventions — Sirolimus; Mycophenolic Acid; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Drug conversion to sirolimus (Active Comparator): Drug conversion to sirolimus: mycophenolate or azathioprine conversion to sirolimus, in a regimen with tacrolimus and prednisone.
  Interventions: Drug: Drug conversion to sirolimus
- Maintenance of the current regimen (Active Comparator): Maintenance of the current regimen: mycophenolate or azathioprine maintenance, in a regimen with tacrolimus and prednisone.
  Interventions: Drug: Maintenance of the current regimen

INTERVENTIONS:
Drug: Drug conversion to sirolimus — Drug conversion to sirolimus: mycophenolate or azathioprine conversion to sirolimus, in a regimen with tacrolimus and prednisone.
  Other Names: Rapamune
  Arms: Drug conversion to sirolimus
Drug: Maintenance of the current regimen — Maintenance of the current regimen: mycophenolate or azathioprine maintenance, in a regimen with tacrolimus and prednisone.
  Other Names: Myfortic; Immuran
  Arms: Maintenance of the current regimen

SUMMARY:
Cytomegalovirus is the most important opportunistic infection after kidney transplant, with increased in mortality, morbidity and higher costs of transplantation. Despite the favorable efficacy (lower acute rejection) results of the most worldwide used regime, tacrolimus, mycophenolate and prednisone, or the investigators local common regimen, tacrolimus, azathioprine and prednisone, this combinations are associated with higher incidence of cytomegalovirus infection, disease and recurrence.

Namely, sirolimus use is associated with decreased risk of cytomegalovirus infection/disease, and there is not a prospective cohort to evaluate the conversion to sirolimus efficacy to decrease the cytomegalovirus infection recurrence.

Given this, the investigators propose a study of their own initiative that attends local needs: evaluate the conversion to sirolimus efficacy in decrease the cytomegalovirus recurrence after kidney transplant.

DETAILED DESCRIPTION:
This protocol is a prospective, randomized, single center, designed to evaluate incidence of cytomegalovirus recurrence infection/disease in two immunosuppressive regimens, after the first episode of cytomegalovirus: (1) conversion of azathioprine or mycophenolate to sirolimus, in a regimen wih low doses tacrolimus and prednisone; ( 2) Maintenance of the current regimen during the first episode of cytomegalovirus infection ( azathioprine or mycophenolate, in combination to tacrolimus or prednisone). Our hypothesis is that conversion from azathioprine or sodium mycophenolate to sirolimus, with low doses of tacrolimus, and prednisone results in lower recurrence of cytomegalovirus infection/disease in kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Adult kidney transplant recipients > 18 y.o.
* Kidney Transplant recipients, after the first episode of cytomegalovirus infection, using the current immunosuppressive regimen: azathioprine or mycophenolate, tacrolimus and prednisone.

Exclusion Criteria:

* Re-transplant;
* Patients with any panel reactive antibody (PRA) equal to or above 50%, class I or class II;
* Acute rejection episode in the last 30 days, or episode > 2A in the Banff criteria;
* GFR (MDRD) < 40 ml/min;
* Proteinuria > 0,5 g/l;
* Hemoglobin < 10 g/l and/or leucocytes < 4000 cels/mm3 and/or platelets < 150.000 cels/mm3;
* Triglycerides > 500 mg/dl with or without use of fibrate;
* Cholesterol total > 300 mg/dl with or without use of statin;
* Hepatic abnormalities;
* Significant periphery edema;
* Pulmonary abnormalities or breast x-ray abnormalities;
* Hyper sensibility to sirolimus formula;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-09; Primary Completion 2019-12 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Cytomegalovirus infection/disease recurrence | One year
  Cytomegalovirus infection/disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Geovana Basso, MD, Principal Investigator — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil; Helio Tedesco Silva Junior, PhD, Study Chair — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil; Claudia Rosso felipe, PhD, Study Chair — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil; Leonardo V. Riella, PhD, Study Chair — Brigham and Women's Hospital, US.; Jose O. Medina Pestana, PhD, Study Chair — Nephrology Division, Hospital do Rim, Federal University of São Paulo, Brazil
Locations (1):
- Hospital do Rim, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Viana LA, Cristelli MP, Basso G, Santos DW, Dantas MTC, Dreige YC, Requiao Moura LR, Nakamura MR, Medina-Pestana J, Tedesco-Silva H. Conversion to mTOR Inhibitor to Reduce the Incidence of Cytomegalovirus Recurrence in Kidney Transplant Recipients Receiving Preemptive Treatment: A Prospective, Randomized Trial. Transplantation. 2023 Aug 1;107(8):1835-1845. doi: 10.1097/TP.0000000000004559. Epub 2023 Jul 20. PMID 37046380